CLINICAL TRIAL: NCT07308561
Title: The Relationship Between Quality of Life, Anxiety Levels, and Attitudes Toward Artificial Intelligence Among Women Undergoing Infertility Treatment
Status: Recruiting | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Güzin Ünlü Suvari, M.Sc., Lecturer, Acibadem University
Other Study IDs: 2025-15/591
Record Dates: First submitted 2025-12-17; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Infertility, Female; Artificial Intelligence; Quality of Life; Anxiety
MeSH Terms: conditions — Infertility, Female; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
Infertility affects approximately one in six individuals worldwide and is associated with significant psychological distress, particularly among women undergoing treatment. Increased anxiety levels are strongly linked to reduced quality of life during the infertility process. With the growing integration of artificial intelligence (AI) into healthcare, AI-based tools are increasingly used in infertility care to support decision-making and patient engagement. While many patients are familiar with AI technologies, individual attitudes toward AI may influence their acceptance and potential psychosocial benefits. This study aims to examine the relationship between attitudes toward artificial intelligence, anxiety levels, and quality of life among women undergoing infertility treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years diagnosed with infertility (primary or secondary infertility).
* Women undergoing infertility treatment and those who have experienced various treatment modalities (IUI, IVF, ICSI).
* Women who voluntarily agree to participate in the study.
* Women who are able to understand and speak Turkish.

Exclusion Criteria:

* Women with diagnosed psychological disorders (e.g., clinical depression, anxiety disorders).
* Women who are not undergoing infertility treatment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18-45 years diagnosed with primary or secondary infertility and currently undergoing infertility treatment (IUI, IVF, or ICSI).
Sampling Method: Non-Probability Sample
Enrollment: 191 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic and Descriptive Information Form | At baseline (one-time assessment at enrollment)
  This form includes 30 items designed to collect data on participants' sociodemographic characteristics, general health status, obstetric and gynecological history, and use of technology and artificial intelligence. It provides a comprehensive background profile of women undergoing infertility treatment.
State-Trait Anxiety Inventory (STAI) - Trait Anxiety Scale | At baseline (one-time assessment at enrollment)
  The Trait Anxiety Scale is used to assess individuals' general and persistent anxiety levels. The scale consists of multiple items rated on a Likert-type format, with total scores ranging from 20 to 80. Higher scores indicate higher levels of anxiety.
General Attitudes Toward Artificial Intelligence Scale | At baseline (one-time assessment at enrollment)
  This scale assesses individuals' positive and negative attitudes toward artificial intelligence using a 5-point Likert-type format. It consists of 20 items, with negatively worded items reverse-coded. Higher total scores reflect more positive attitudes toward artificial intelligence.
Fertility Quality of Life Scale (FertiQol) - Core Module | At baseline (one-time assessment at enrollment)
  The Fertility Quality of Life Scale evaluates quality of life in individuals experiencing fertility problems. The core module assesses emotional, mind-body, relational, and social dimensions of quality of life using a Likert-type response format. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Health Group, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared due to privacy concerns and the sensitive nature of maternal and infant health information. However, anonymized data may be made available upon reasonable request to the corresponding author after publication of the study results.

REFERENCES:
- [Background] European Society of Human Reproduction and Embryology (ESHRE). (2024, April). Factsheet on infertility - prevalence, treatment and fertility decline in Europe. ESHRE. https://www.eshre.eu
- [Background] Shi Z, Zheng Y, Zhu X, Mao Z, Nie H, Chen G, Li S. Understanding health-related quality of life in Chinese infertility patients: a qualitative study. Qual Life Res. 2025 Nov;34(11):3105-3119. doi: 10.1007/s11136-025-04066-y. Epub 2025 Sep 13. PMID 40944797
- [Background] Simionescu G, Doroftei B, Maftei R, Obreja BE, Anton E, Grab D, Ilea C, Anton C. The complex relationship between infertility and psychological distress (Review). Exp Ther Med. 2021 Apr;21(4):306. doi: 10.3892/etm.2021.9737. Epub 2021 Feb 1. PMID 33717249
- [Background] Song D, Li X, Yang M, Wang N, Zhao Y, Diao S, Zhang X, Gou X, Zhu X. Fertility quality of life (FertiQoL) among Chinese women undergoing frozen embryo transfer. BMC Womens Health. 2021 Apr 24;21(1):177. doi: 10.1186/s12905-021-01325-1. PMID 33894750
- [Background] Gameiro S, Boivin J, Dancet E, de Klerk C, Emery M, Lewis-Jones C, Thorn P, Van den Broeck U, Venetis C, Verhaak CM, Wischmann T, Vermeulen N. ESHRE guideline: routine psychosocial care in infertility and medically assisted reproduction-a guide for fertility staff. Hum Reprod. 2015 Nov;30(11):2476-85. doi: 10.1093/humrep/dev177. Epub 2015 Sep 7. PMID 26345684
- [Background] Cromack SC, Lew AM, Bazzetta SE, Xu S, Walter JR. The perception of artificial intelligence and infertility care among patients undergoing fertility treatment. J Assist Reprod Genet. 2025 Mar;42(3):855-863. doi: 10.1007/s10815-024-03382-5. Epub 2025 Jan 7. PMID 39776390
- [Background] Medenica S, Zivanovic D, Batkoska L, Marinelli S, Basile G, Perino A, Cucinella G, Gullo G, Zaami S. The Future Is Coming: Artificial Intelligence in the Treatment of Infertility Could Improve Assisted Reproduction Outcomes-The Value of Regulatory Frameworks. Diagnostics (Basel). 2022 Nov 28;12(12):2979. doi: 10.3390/diagnostics12122979. PMID 36552986
- [Background] Sarshoori, A. A., Mostafavi, M., Heidarpoor, S., & Chekeni, A. M. (2024). Role of Artificial Intelligence in Infertility Screening and Treatment: A Systematic Review. Iranian Biomedical Journal, 28, 253.
- [Background] Lee, C., Chae, H. J., Kim, H. M., Lee, H., Choi, S., & Min, H. S. (2024). Enhancing infertility care with a ChatGPT-based chatbot: integrating clinical and community insights for improved patient support. Fertility and Sterility, 122(4), e141-e142.
- [Background] Méndez-Suárez, M., Delbello, L., de Vega de Unceta, A., & Ortega Larrea, A. L. (2024). Factors affecting consumers' attitudes towards artificial intelligence. Journal of Promotion Management, 30(7), 1141-1158.
- [Background] Mendizabal-Ruiz G, Paredes O, Borrayo E, Chavez-Badiola A. FERTILITY CARE IN LOW- AND MIDDLE- INCOME COUNTRIES: The future use of AI to improve accessibility of assisted reproductive technology in low- and middle-income countries. Reprod Fertil. 2025 Aug 14;6(3):e240077. doi: 10.1530/RAF-24-0077. Print 2025 Jul 1. PMID 40736784
- [Background] Massarotti C, Gentile G, Ferreccio C, Scaruffi P, Remorgida V, Anserini P. Impact of infertility and infertility treatments on quality of life and levels of anxiety and depression in women undergoing in vitro fertilization. Gynecol Endocrinol. 2019 Jun;35(6):485-489. doi: 10.1080/09513590.2018.1540575. Epub 2019 Jan 7. PMID 30612477
- [Background] Braverman AM, Davoudian T, Levin IK, Bocage A, Wodoslawsky S. Depression, anxiety, quality of life, and infertility: a global lens on the last decade of research. Fertil Steril. 2024 Mar;121(3):379-383. doi: 10.1016/j.fertnstert.2024.01.013. Epub 2024 Jan 13. PMID 38224730
- [Background] Kaya, F., Aydin, F., Schepman, A., Rodway, P., Yetişensoy, O., & Demir Kaya, M. (2022). The roles of personality traits, AI anxiety, and demographic factors in attitudes towards artificial intelligence. International Journal of Human-Computer Interaction. https://doi.org/10.1080/10447318.2022.2151730
- [Background] Schepman A, Rodway P. Initial validation of the general attitudes towards Artificial Intelligence Scale. Comput Hum Behav Rep. 2020 Jan-Jul;1:100014. doi: 10.1016/j.chbr.2020.100014. Epub 2020 May 18. PMID 34235291
- [Background] Schepman, A. & Rodway, P. (2022). The General Attitudes towards Artificial Intelligence Scale (GAAIS): Confirmatory Validation and Associations with Personality, Corporate Distrust, and General Trust. International Journal of Human-Computer Interaction https://doi.org/10.1080/10447318.2022.2085400